CLINICAL TRIAL: NCT04432012
Title: Comparison of Perioperative Intravenous vs Periarticular Dexamethasone vs no Steroid Supplementation in Terms of Post-operative Pain, Function, Nausea, Hospitalization Length, and Risk of Complications in Patients Undergoing Primary Total Knee Arthroplasty for Knee Osteoarthritis - A Randomized Controlled Trial Clinical Study Protocol
Brief Title: A Study to Compare Different Ways of Steroid Administration After Total Knee Implantation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Christian Candrian (Other)
Responsible Party: Sponsor-Investigator, Christian Candrian, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORL-ORT-013
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Total Knee Replacement
Keywords: Knee; surgery; replacement; arthroplasty
MeSH Terms: interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The present study will be double blinded: both participants and assessor will be blinded to the assigned treatment. Only the surgeons and the anaesthetists taking part to surgery will be aware of the group to which the patient was assigned but they will not take part to the follow-up visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- arm-A Intra-venous dexamethasone (Experimental): 9 mg of Intra-venous dexamethasone
  Interventions: Drug: Dexamethasone Sodium Phosphate 4 mg/ml intravenous
- arm-B intra-articular dexamethasone (Experimental): 9 mg of intra-articular dexamethasone
  Interventions: Drug: Dexamethasone Sodium Phosphate 4 mg/ml intra-articular
- arm-C routine (No Intervention): No steroid supplementation or other drugs will be added to the routinely performed anaesthesia protocol in the control group

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate 4 mg/ml intravenous — Perioperative intravenous injection of 3 ml of solution (9mg of dexamethasone)
  Other Names: Mephameson
  Arms: arm-A Intra-venous dexamethasone
Drug: Dexamethasone Sodium Phosphate 4 mg/ml intra-articular — Perioperative intra-articular injection of 3 ml of solution (9mg of dexamethasone)
  Other Names: Mephameson
  Arms: arm-B intra-articular dexamethasone

SUMMARY:
We are going to evaluate the difference between perioperative intravenous steroid supplementation, perioperative periarticular steroid supplementation, and standard anaesthesia protocols. We'll evaluate the outcome of patients with knee osteoarthritis who are undergoing Total Knee Arthroplasty to understand which of the three treatments give more benefits to the patient.

DETAILED DESCRIPTION:
A total of 159 patients will be needed (53 patients per arm, 3 arms in total). Dexamethasone (brand name: Mephameson) is the steroid drug that we perioperative administer in two different ways: intra-venous (IV) dexamethasone (9mg) in arm-A, intra-articular (IA) dexamethasone (9mg) in arm-B. No steroid supplementation will be provided in the control group (arm-C).

The primary objective of the study is to compare the effect on post-operative pain of I.V. and I.A. perioperative dexamethasone supplementation for total knee arthroplasty (TKA).

The secondary objectives of the studies will be the comparison between I.V. and I.A. peri-operative dexamethasone supplementation in terms of post-operative pain and function, opioids and analgesic drugs consumption, knee range of motion, systemic inflammatory response, time to mobilisation, length of stay, and patient satisfaction.

Moreover, both I.V. and I.A. steroid supplementation protocols will be compared to routine analgesia protocol (no steroid supplementation group) in order to document their advantages over the absence of steroid supplementation.

The safety of I.V. and I.A. peri-operative dexamethasone will be evaluated and compared recording all the steroid supplementation related complications. In particular, the risk of hyperglycaemia-related complications and post-operative infections will be documented. The safety of both I.V. and I.A. steroid supplementation protocols will be verified comparing them to the no-treatment group in terms of incidence of complications.

Overall study duration will be 12 years: 2 years to enroll all the patients and 10 years to complete the last follow-up. Primary data analysis is planned after the completion of the 1-year follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary TKA at the Ospedale Regionale di Lugano.
* Patients with a BMI >18.5 and <35.
* Patients able to provide informed consent and follow all the study procedures as indicated by the protocol.
* Informed Consent as documented by signature (Appendix Informed Consent Form).

Exclusion Criteria:

* Contraindications to steroids.
* Revision TKA.
* Active steroid therapy.
* Women who are pregnant or breast feeding.
* Presence of other clinically significant concomitant disease states (ASA IV).
* Uncontrolled diabetes mellitus
* Known or suspected non-compliance, drug or alcohol abuse.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Previous enrolment into the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2033-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean daily pain at rest during the first 3 days on a 0-10 numeric rating scale | 3 days after surgery
  Mean daily pain at rest during the first 3 days reported on a 0-10 numeric rating scale (NRS) by the patients.
  The 0-10 NRS consists in a single 11-point numeric scale, with 0 indicating no pain and 10 reflecting the worst possible pain.

SECONDARY OUTCOMES:
Post-operative knee pain during the first 6 weeks after surgery on a 0-10 numeric rating scale | 6 weeks after surgery
  Pain reported on 0-10 numeric rating scale (NRS) during the first 6 weeks and documented with a mobile application (developed at our Institution) that will ask the patients to report pain twice a day (once in the morning, once in the evening). Comparison will be performed in terms of mean daily pain during the first 6 weeks and mean daily pain during every single week.
  The 0-10 NRS consists in a single 11-point numeric scale, with 0 indicating no pain and 10 reflecting the worst possible pain.
Post-operative knee pain during the first 10 years after surgery | 10 years
  reported on 0-10 NRS at 3, 6, 12, 24, 60 and 120 months using a questionnaire. The 0-10 NRS consists in a single 11-point numeric scale, with 0 indicating no pain and 10 reflecting the worst possible pain.
Post-operative function during the first 6 weeks after surgery | 6 weeks
  reported on 0-10 NRS 8see above) during the first 6 weeks, documented with a mobile application developed by our institution that will ask the patients to report pain twice a day (once in the morning, once in the evening). Comparison will be performed in terms of mean daily pain during the first 6 weeks and mean daily pain during every single week. Furthermore, pain trajectories will be created.
  The 0-10 NRS consists in a single 11-point numeric scale, with 0 indicating the worst possible function and 10 reflecting the best possible function.
Post-operative knee function during the first 10 years after surgery | 10 years
  reported on 0-10 NRS at 3, 6, 12, 24, 60 and 120 months using a questionnaire. The 0-10 NRS consists in a single 11-point numeric scale, with 0 indicating the worst possible function and 10 reflecting the best possible function.
Post-operative knee outcome on Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 10 years
  Questionnaire at 2 and 6 weeks, and at 3, 6, 12, 24, 60 and 120 months. The WOMAC questionnaire is composed of 3 sub-scores that evaluate pain (5 questions, 0-20 points), stiffness (2 questions, 0-8 points), and function (17 questions, 0-68 points) and is a validated patient-reported outcome measure (PROM) to evaluate knee osteoarthritis.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Knee conditions on Knee society score (KSS) | 10 years
  Questionnaire at 2 and 6 weeks, and at 3, 6, 12, 24, 60 and 120 months. The original KSS has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
Quality of pain on PainDETECT questionnaire | 10 years
  Questionnaire at 2 and 6 weeks, and at 3, 6, 12, 24, 60 and 120 months. PainDETECT consists of seven questions that address the quality of pain symptoms; it is completed by the patient and no physical examination is required. A score ≤12 indicates that pain is unlikely to have a neuropathic component (< 15%), while a score of ≥19 suggests that pain is likely to have a neuropathic component (> 90%). An intermediate score (≥13, ≤18) indicates a possible neuropathic component .
Patient satisfaction: numeric rating scale (NRS) | 10 years
  Patient satisfaction reported on 0-10 numeric rating scale (NRS) at 3, 6, 12, 24, 60 and 120 months using a questionnaire.
  The 0-10 NRS consists in a single 11-point numeric scale, with 0 indicating that patient is not satisfied at all and 10 reflecting that patient is totally satisfied.
Post-operative nausea incidence | During Hospitalization, approximately 3 days
  incidence (on a 0-10 NRS) of nausea will be evaluated in the first post-operative days.
  The 0-10 NRS consists in a single 11-point numeric scale, with 0 indicating no nausea and 10 reflecting the maximum intensity of nausea.
Post-operative nausea intensity | During Hospitalization, approximately 3 days
  intensity (on a 0-10 NRS) of nausea will be evaluated in the first post-operative days.
  The 0-10 NRS consists in a single 11-point numeric scale, with 0 indicating no nausea and 10 reflecting the maximum intensity of nausea.
Post-operative opioids and analgesic drugs consumption | During Hospitalization, approximately 3 days
  Medication Quantification Scale (MQS) score will be used to evaluate analgesic drug consumption.
  Medication Quantification Scale (MQS) scor is calculated for each medication by taking a consensus-based detriment weight for a given pharmacologic class and multiplying it by a score for dosage. The calculated values for each medication are then summed for a total MQS score. The score can provide a useful point measure of medication usage for any pain medication regimen.
Post-operative C-Reactive Protein (CRP) | every days 3 days from surgery
  Hematic C-Reactive Protein in mg/L will be evaluated as index of post-operative inflammatory response.
Post-operative erythrocyte sedimentation rate (ESR) | every days 3 days from surgery
  Erythrocyte sedimentation rate (mm/h) will be evaluated as index of post-operative inflammatory response.
Time from surgery to first mobilization | During Hospitalization, approximately 1 days
Time needed for climbing stairs the first time | approximately 1 week
Length of hospital stay | approximately 1 week

OTHER OUTCOMES:
Number of patients with treatment-related adverse events | 10 years
  The safety of I.V. and I.A. dexamethasone supplementation will be evaluated in terms of: rate of serious adverse events related to steroid supplementation, rate of prosthetic joint infections, rate of wound infections, rate of wound healing problems.
  Furthermore, glycaemia will be evaluated daily during the first three days after surgery.
  To delineate a complete safety profile of dexamethasone supplementation, all treatment related adverse events will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Candrian, MD, Prof., Principal Investigator — EOC
Locations (1):
- Ospedale Regionale di Lugano Civico e Italiano, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No
not foreseen